CLINICAL TRIAL: NCT02635880
Title: A Clinical Evaluation of a Novel Multi-Wavelength Laser for Benign Pigmented Lesion Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-15-EN08
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2016-01

CONDITIONS: Pigmented Skin Lesion of Suspected Benign Nature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Investigational Enlighten Device (Experimental): Laser treatment for removal of benign pigmented lesions (BPLs) with Nd:YAG dual-wavelength, dual-pulse duration laser.
  Interventions: Device: Investigational Enlighten Device

INTERVENTIONS:
Device: Investigational Enlighten Device — Up to 3 laser treatments, spaced 4 to 6 weeks apart

SUMMARY:
To evaluate the safety and efficacy of an investigational version of the Cutera enlightenTM laser that offers multiple wavelengths for removal of benign pigmented lesions.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate the safety and efficacy of an investigational version of the Cutera enlightenTM laser for benign pigmented lesion (BPL) removal. Currently, the enlightenTM laser offers two wavelengths: 532nm KTP and 1064nm Nd:YAG. The version of the laser under investigation allows the user to choose from a range of wavelengths.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - III (Appendix 3).
* Clinical diagnosis of benign pigmented lesions located on the hand, body or face.
* Presence of 5 or more benign pigmented lesions in the treatment area, ranging in diameter from 2 to 8 mm.
* Has not used any prescription or over-the-counter topical creams (such as hydroquinone, retinoids or corticosteroids) in the designated treatment area within 4 weeks of enrollment in the study and is willing to refrain from use for the duration of the study.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Wiling to cover treated area or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and every day for the duration of the study, including the follow-up period.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) for the treatment of BPL during the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study.

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as chemical peel, laser or light-based procedure, or surgery.
* Presence of pre-malignant or malignant lesion in the treatment area (such as, but not limited to pigmented actinic keratosis, lentigo maligna or lentigo maligna melanoma) or history of a pre-malignant or malignant lesion in the treatment area.
* Shows signs of actinic bronzing and/or excessively tanned in areas to be treated, and unable or unlikely to refrain from tanning during the study (for example, subject's occupation requires regular sun exposure).
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid or isotretinoin within 12 months of study participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Moldre, NP, Principal Investigator — Cutera Inc.
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healty Evaluation of Clinical Study: Laser treatment for removal of benign pigmented lesions (BPLs) with Nd:YAG dual-wavelength, dual-pulse duration laser.
Period: Overall Study
Arm/Group | Healty Evaluation of Clinical Study
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Group: The following types of benign pigmented lesions will be treated in this study: (1) lentigines (solar or senile); (2) ephelides (freckles); and (3) seborrheic keratosis.
Arm/Group | Baseline Group
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Change of Treated Lesions
Description: Degree of change in treated lesions at 6 weeks post-final treatment as assessed using the Global Aesthetic Improvement Scale (GAIS) with a scoring of 0 - for no change, 1 - Mild Improvement, 2 - Moderate Improvement, 3 - Significant Improvement, 4 - Very SIgnificant Improvement.
Time Frame: Baseline and 6 weeks post-final treatment
Measure: Number; unit: % of participants
Arm/Group | Investigational Enlighten Device
Number analyzed (Participants) | 32
% of participants
  Complete Improvement | 44
  Moderate Improvement | 44
  Mild Improvement | 13

2. Secondary Outcome: Percentage of Particpant Satisfaction of Improvement in Treated Lesions by the Subject
Description: Degree of improvement in treated lesions at 6 weeks post-final treatment as assessed by the subject through a customized subject satisfaction survey. Survey was based upon a scoring 0 - Extremely Unsatisfied, 1 - Unsatisfied, 2 - Neutral, 3- Satisfied, 4 - Extremely Satisfied.
Time Frame: 6 weeks post-final treatment
Measure: Number; unit: % of participants
Arm/Group | Investigational Enlighten Device
Number analyzed (Participants) | 32
% of participants
  Neutral | 6
  Satisfied | 38
  Extremely Satisified | 56

ADVERSE EVENTS:
Arm/Group | Investigational Enlighten Device
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No